CLINICAL TRIAL: NCT02745314
Title: Effectiveness of Physical Frailty Measurement to Determine the Outcome of Elderly Patients With Severe Symptomatic Aortic Stenosis
Brief Title: Frailty and Mortality in Older Old With Severe Aortic Stenosis
Acronym: SAS-frailty
Status: Completed | Type: Observational
Sponsor: Hospital de Meixoeiro (Other Government)
Responsible Party: Principal Investigator, Carlos RodrÃ-guez Pascual, MD, PhD, Hospital de Meixoeiro
Other Study IDs: HMeixoeiro
Record Dates: First submitted 2016-04-16; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis, Frailty, Elderly, moertality
MeSH Terms: conditions — Aortic Valve Stenosis; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- >74 years: Older than 74 year-old patients
  Interventions: Other: Frailty measurement; Other: Comprehensive Geriatric Assessment

INTERVENTIONS:
Other: Frailty measurement — Frailty measurement under Fried at el criteria
Other: Comprehensive Geriatric Assessment — Multidimensional Geriatric Assessment

SUMMARY:
BACKGROUND.- The frailty syndrome (FS) associates an increase in morbidity and mortality in the elderly patient. When severe and symptomatic, aortic stenosis (AS) is a disease with poor prognosis, the most frequent cause of heart surgery in the elderly and associates high health costs. No variables have been identified as determinants of morbidity and mortality of these patients and there are not algorithms developed for treatment decision-making in this particular population. The FS as a functional reserve indicator could be a prognostic and interventional treatment tolerance marker, and should be included in the selection of patients for surgical treatment. The FS and cardiovascular disease (CVD) share biological substrates among which an inflammatory state associates poor prognosis.

OBJECTIVES .- To evaluate the effectiveness of the diagnosis of FS to characterize the prognosis of elderly patients with severe symptomatic AS representative of clinical practice. In addition, to examine the contribution of an inflammatory state to the relationship of FS with the prognosis of severe, symptomatic AS.

METHODS .- Prospective study during 12 months of 200 patients > 74 years old with severe symptomatic AS. During the index visit the main clinical characteristics will be recorded and in addition we will perform a comprehensive geriatric assessment, FS assessmet according to Fried et al criteria (strength, walking speed, physical activity, fatigue, unintentional weight loss) and determination of inflammatory markers (C-reactive protein and interleukin-6). During follow-up, measures of functional impairment (basic and instrumental activities of daily living, walking speed and timed set up & go test), hospitalizations, death and quality of life will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis
* 75 years or older
* Ambulatory

Exclusion Criteria:

* Life expectancy lower than one year
* Severe cognitive decline
* Previous intervention on aortic valve

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older than 74 year-old patients with symptomatic severe aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mortality | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Meixoeiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No
Not initially considered but open to external collaboration

REFERENCES:
- [Derived] Pinon M, Paredes E, Acuna B, Raposeiras S, Casquero E, Ferrero A, Torres I, Legarra JJ, Pradas G, Barreiro-Morandeira F, Rodriguez-Pascual C. Frailty, disability and comorbidity: different domains lead to different effects after surgical aortic valve replacement in elderly patients. Interact Cardiovasc Thorac Surg. 2019 Sep 1;29(3):371-377. doi: 10.1093/icvts/ivz093. PMID 31220291